CLINICAL TRIAL: NCT02776683
Title: A Single Arm, Open-label, Multicenter, Multinational, Safety and Efficacy Phase IIIb Trial of BI 695502 Plus mFOLFOX6 in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Open-label, Single Arm Trial of BI 695502 in Patients With Previously Untreated Metastatic Colorectal Cancer
Acronym: INVICTAN®-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1302.3; 2015-003718-25 (EudraCT Number)
Record Dates: First submitted 2016-05-17; First posted 2016-05-18 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

ARMS (1):
- All patients (Experimental)
  Interventions: Drug: BI 695502; Drug: Avastin

INTERVENTIONS:
Drug: BI 695502
Drug: Avastin

SUMMARY:
The objective of this trial is to evaluate the safety and tolerability of BI 695502 in combination with leucovorin/5-fluorouracil/oxaliplatin (mFOLFOX6) and as maintenance therapy (when applicable). As well as to evaluate the following efficacy parameters: Progression-free survival (PFS), objective response rate (proportion of patients with complete response [CR] plus partial response [PR]), overall survival (OS), duration of response (DOR), time to progression (TTP).

ELIGIBILITY:
Inclusion criteria:

* Males and females aged >=18 years (for Japan only: Age >=20 years at time of signing Informed Consent Form) with histologically confirmed metastatic colorectal cancer (mCRC).
* Metastatic disease not amenable to surgical curative treatment and eligible to receive therapy with mFOLFOX6 (Leucovorin/5-Fluorouracil/Oxaliplatin) + bevacizumab.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Adequate hepatic, renal and bone marrow function.
* Further inclusion criteria apply.

Exclusion criteria:

* Prior systemic therapy for metastatic disease
* Prior therapy with monoclonal antibodies or small molecule inhibitors against Vascular endothelial growth factor (VEGF) or VEGF receptors, including Avastin® or Avastin® biosimilar
* Previous malignancy other than Colorectal cancer (CRC) in the last 5 years except for basal cell cancer of the skin or pre-invasive cancer of the cervix
* Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 6 weeks prior to start of study treatment
* Any unresolved toxicity > Common Toxicity Criteria Grade 1 (except alopecia) from previous anticancer therapy (including radiotherapy)
* History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
* A thrombotic or hemorrhagic event <=6 months prior to screening (includes hemoptysis, Gastrointestinal (GI) bleeding, hematemesis, central nervous system hemorrhage, epistaxis, vaginal bleeding, cerebral infarction, transient ischemic attacks, myocardial infarction, angina, and coronary artery disease)
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (46):
- United States (25):
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - The Oncology Institute of Hope and Innovation, Anaheim, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Ashland Bellefonte Cancer Center, Ashland, Kentucky
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Aultman Hospital, Canton, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Northwest Cancer Specialists PC, Portland, Oregon
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Texas Oncology, P.A., Abilene, Texas
  - Texas Oncology, PA,, Amarillo, Texas
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, P.A., Flower Mound, Texas
  - Texas Oncology, P.A., Garland, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Texas Oncology, P.A., McAllen, Texas
  - Texas Oncology, PA, Mesquite, Texas
  - Texas Oncology-San Antonio Northeast, San Antonio, Texas
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - Tyler Hematology-Oncology, PA, Tyler, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - Texas Oncology, P.A., Deke Slayton Cancer Center, Webster, Texas
  - Virginia Cancer Institute, Richmond, Virginia
- Japan (7):
  - Chiba Cancer Center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Ehime, Matsuyama
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Japan Organization of Occupational Health and Safety Kansai Rosai Hospital, Hyogo, Amagasaki
  - Kagawa University Hospital, Kagawa, Kita-gun
  - Osaka University Hospital, Osaka, Suita
  - Jananese Foundation for Cancer Research, Tokyo, Koto-ku
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Clínico de Valencia, Valencia
- Ukraine (11):
  - CI Chernivtsi RC Oncological Dispensary Bukovinian SMU, Chernivtsi
  - Munic.Instit."City Clin.Hosp.#4" of Dnipro City Council, Dnipropetrovsk
  - Regional Clinical Oncological Dispensary, Ivano-Frankivsk, Ivano-Frankivsk
  - CI of PH Kharkiv CCH #2, Kharkiv
  - Treatment-Diagnostic CTR of Private Enterprise, Kirovohrad, Kirovohrad
  - CI Kryvyi Rih Oncological Dispensary of DRC, Kryvyi Rih, Dnipropetrovsk
  - National Institute of Cancer, Kyiv
  - CI of LRC Lviv Onco.Reg.Treat.&Diag.Cent., Lviv
  - Poltava Regional Clinical Oncological Dispensary, Poltava, Poltava
  - Sumy Regional Oncology Center, Sumy
  - Vinnytsia Regional Clinical Oncological Dispensary, Vinnytsia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was Phase IIIb, open-label, multicenter, multinational, single-arm trial. Patients with previously untreated metastatic colorectal cancer (mCRC) were enrolled. From 21December2017, Sponsor recommended that patients should be switched from BI 695502 to the reference product Avastin® as soon as it was available at the respective clinical site.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that they (the patient) met all strictly implemented inclusion/exclusion criteria. Patients were not to be randomised to trial treatment if any one of the specific entry criteria were violated.
Groups:
- BI 695502: All patients were to receive BI 695502 (5 milligrams per kilogram [mg/kg]) solution for intravenous (i.v.) infusion in combination with mFOLFOX6 chemotherapy every 2 weeks. Patients were to continue to receive treatment during the pre-switch period until disease progression, death, unacceptable toxicity, or the end of the trial, whichever occurred earlier. Based on patient tolerability, at least 8 cycles of mFOLFOX6 were to be given to all patients.
- BI 695502 to Avastin®: At the switch visit, patients were to be switched from BI 695502 to Avastin®. Post-switch, patients were to receive Avastin® (5 mg/kg) solution for i.v. infusion in combination with mFOLFOX6 chemotherapy every 2 weeks. Patients were to continue to receive treatment until disease progression, death, unacceptable toxicity, or the end of the trial, whichever occurred earlier.
Period: Pre-switch Period
Arm/Group | BI 695502 | BI 695502 to Avastin®
Started (Only the BI 695502 arm was applicable for Period 1) | 123 (Assigned to trial medication or enrolled/treated) | 0
Completed | 43 (Entered into Switch Set) | 0
Not Completed | 80 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 21 | 0
Not completed — Withdrawal by Subject | 9 | 0
Not completed — Physician Decision | 7 | 0
Not completed — Progressive disease | 39 | 0
Not completed — Other than listed | 3 | 0
Period: Post-switch Period
Arm/Group | BI 695502 | BI 695502 to Avastin®
Started (Only the BI 695502 to Avastin arm was applicable to Period 2) | 0 | 43 (Entered into Switch Set)
Completed | 0 | 0
Not Completed | 0 | 43
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Progressive disease | 0 | 20
Not completed — Other than listed | 0 | 15

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS contained all participants who signed informed consent and who received at least one dose of trial medication.
Arm/Group | BI 695502
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 33
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 82
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Treatment-Emergent Adverse Events (TEAEs) in the Specified Categories Selected for Primary Endpoint Assessment
Description: The primary safety endpoint of the trial was patients with any of the following selected adverse events (AEs):
  * Infusion reactions (anaphylactic/hypersensitivity/infusion-related reactions),
  * Thromboembolic events (arterial or venous),
  * Gastrointestinal perforations,
  * Hypertension,
  * Proteinuria,
  * Pulmonary hemorrhage
  * All hemorrhages (including pulmonary hemorrhages)
  * Wound-healing complications/abscess/fistulas
  * Posterior reversible encephalopathy syndrome
  * Ovarian failure. All AEs with an onset between start of treatment and end of the residual effect period (REP), a period of 18 weeks after the last dose of trial medication were considered for the primary safety analysis. Confidence interval was calculated using Wilson score method.
Time Frame: From baseline up to 18 weeks after the last dose of trial medication prior to the Switch Visit. Maximum duration of up to 32 treatment cycles + safety follow up (up to 82 weeks overall).
Population: Treated set (TS): The TS contained all patients who signed informed consent and who received at least one dose of trial medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | BI 695502
Number analyzed (Participants) | 123
Percentage of participants (%)
  Patients with any of the selected AEs | 58.5 [49.70 to 66.86]
  Infusion reactions | 18.7 [12.80 to 26.50]
  Thromboembolic events | 12.2 [7.53 to 19.15]
  Gastrointestinal perforations | 2.4 [0.83 to 6.93]
  Hypertension | 28.5 [21.23 to 36.99]
  Proteinuria | 9.8 [5.67 to 16.28]
  Pulmonary Haemorrhage | 0.00 [0.00 to 3.03]
  Hemorrhages | 22.80 [16.25 to 30.93]
  Wound-healing complications | 1.6 [0.45 to 5.74]
  Reversible Encephalopathy Syndrome | 0.0 [0.00 to 3.03]
  Ovarian failure | 0.00 [0.00 to 6.53]

2. Secondary Outcome: Duration of Response (DOR) as Assessed by Central Imaging Review
Description: DOR was the time from first documented Complete Response (CR) (CR is disappearance of all target lesions) or Partial Response (PR) (PR is at least a 30% decrease in the sum of diameters (SoD) of target lesions taking as reference the baseline sum diameters) until time of progression as assessed by central imaging review per Response evaluation criteria in solid tumors (RECIST) 1.1. RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize") or worsen ("progress") during treatment. DOR was calculated using the Kaplan-Meier technique. Confidence interval was calculated based on the Brookmeyer and Crowley method.
Time Frame: Tumor scans were performed at baseline then every ~8 weeks up to 34 weeks, then every ~12 weeks thereafter until confirmed disease progression. Analysis performed for the pre-switch period only; maximum duration of up to 32 treatment cycles (64 weeks).
Population: TS: The TS contained all patients who signed informed consent and who received at least one dose of trial medication. Only patients with complete or partial objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502
Number analyzed (Participants) | 77
Months | 9.1 [7.3 to NA] — The upper limit confidence interval was not determined as it was not reached

3. Secondary Outcome: Time to Progression (TTP) as Assessed by Central Imaging Review
Description: TTP was defined as the time from first administration of trial medication to the date of tumor progression as assessed by central imaging review per RECIST 1.1 (RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize") or worsen ("progress") during treatment.). TTP was calculated using the Kaplan-Meier technique. Confidence interval was calculated based on the Brookmeyer and Crowley method.
Time Frame: as for outcome 2
Population: TS: The TS contained all patients who signed informed consent and who received at least one dose of trial medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502
Number analyzed (Participants) | 123
Months | 11.1 [9.5 to 12.9]

4. Secondary Outcome: Objective Response (OR) Rate as Assessed by Central Imaging Review
Description: OR rate was defined as the percentage of patients who achieved at least one visit response of CR (CR is disappearance of all target lesions) or PR (PR is at least a 30% decrease in the sum of diameters (SoD) of target lesions taking as reference the baseline sum diameters) after the start of treatment. The response criteria evaluation was carried out according to RECIST 1.1. RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize") or worsen ("progress") during treatment. Confidence interval was calculated using Wilson score method. The definition for OR (CR/PR) extends until disease progression/ death/ unacceptable toxicity/ end of the trial, whichever occurred earlier. However for "Duration of response" this censoring does not apply. Hence the apparent discrepancy.
  OR = CR + PR.
Time Frame: as for outcome 2
Population: TS: The TS contained all patients who signed informed consent and who received at least one dose of trial medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BI 695502
Number analyzed (Participants) | 123
Percentage of participants | 61.0 [52.1 to 69.1]

5. Secondary Outcome: Overall Survival (OS) Time
Description: OS was defined as the time from first administration of trial medication until death from any cause. OS was calculated using the Kaplan-Meier technique. Confidence interval was calculated based on the Brookmeyer and Crowley method.
Time Frame: From date of first dose of trial medication until last date of trial medication + 18 weeks (REP), up to a maximum of 32 treatment cycles + safety follow up (up to 82 weeks overall).
Population: TS: The TS contained all patients who signed informed consent and who received at least one dose of trial medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502
Number analyzed (Participants) | 123
Months | 19.4 [16.7 to 21.1]

6. Secondary Outcome: Progression-Free Survival (PFS) Time as Assessed by Central Imaging Review
Description: PFS was defined as the time from first administration of trial medication until disease progression as assessed by central imaging review or death due to any cause. Disease progression was assessed according to RECIST 1.1. RECIST is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize") or worsen ("progress") during treatment. Progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. PFS was calculated using the Kaplan-Meier technique. Confidence interval was calculated based on the Brookmeyer and Crowley method.
Time Frame: as for outcome 2
Population: TS: The TS contained all patients who signed informed consent and who received at least one dose of trial medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BI 695502
Number analyzed (Participants) | 123
Months | 10.5 [9.4 to 11.8]

ADVERSE EVENTS:
Time Frame: From date of first dose of trial medication until last date of trial medication + 18 weeks (REP), up to a maximum of 32 treatment cycles + safety follow up (up to 82 weeks overall).
Description: All-Cause mortality is defined as death due to any cause (including disease progression) and is reported for the overall study period, including both the pre-switch period for BI 695502 treatment and post-switch period for Avastin® treatment. Serious and other (non-serious) data is based on on-treatment adverse events.
Arm/Group | BI 695502
All-Cause Mortality (participants affected / at risk) | 41/123
Serious Adverse Events (participants affected / at risk) | 33/123
Other Adverse Events (participants affected / at risk) | 118/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695502 (N=123)
Sepsis (Infections and infestations) | 2
Bacterial sepsis (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Hypersplenism (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cervical radiculopathy (Nervous system disorders) | 1
Myelopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Accelerated hypertension (Vascular disorders) | 1
Brachiocephalic vein thrombosis (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Abdominal hernia (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal haematoma (Renal and urinary disorders) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695502 (N=123)
Urinary tract infection (Infections and infestations) | 8
Neutropenia (Blood and lymphatic system disorders) | 32
Anaemia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Leukopenia (Blood and lymphatic system disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 26
Hypokalaemia (Metabolism and nutrition disorders) | 10
Insomnia (Psychiatric disorders) | 9
Peripheral sensory neuropathy (Nervous system disorders) | 44
Neuropathy peripheral (Nervous system disorders) | 21
Dysgeusia (Nervous system disorders) | 18
Headache (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 8
Neurotoxicity (Nervous system disorders) | 7
Hypertension (Vascular disorders) | 34
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Nausea (Gastrointestinal disorders) | 57
Diarrhoea (Gastrointestinal disorders) | 41
Stomatitis (Gastrointestinal disorders) | 37
Constipation (Gastrointestinal disorders) | 27
Vomiting (Gastrointestinal disorders) | 19
Abdominal pain (Gastrointestinal disorders) | 17
Abdominal pain upper (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 16
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Proteinuria (Renal and urinary disorders) | 11
Fatigue (General disorders) | 45
Pyrexia (General disorders) | 17
Malaise (General disorders) | 10
Asthenia (General disorders) | 9
Neutrophil count decreased (Investigations) | 25
Platelet count decreased (Investigations) | 18
Weight decreased (Investigations) | 18
White blood cell count decreased (Investigations) | 18
Gamma-glutamyltransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 7
Weight increased (Investigations) | 7

LIMITATIONS AND CAVEATS:
From 21 December 2017, the Sponsor recommended for patients to be switched from BI 695502 to Avastin®. The main analyses for reporting primary and secondary endpoints was clarified as the pre-switch period (i.e., all receiving BI 695502).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT02776683/SAP_000.pdf
  • Study Protocol (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02776683/Prot_001.pdf